CLINICAL TRIAL: NCT00439634
Title: A 24-Week, Multicenter, Double-Blind, Randomized, Parallel-Group, Dose Ranging Study of the Efficacy and Safety of 3 Oral Doses of AVE1625 and Placebo on Top of Either Olanzapine, Risperidone/Paliperidone, Quetiapine or Aripiprazole in the Treatment of Cognitive Impairment in Schizophrenia.
Brief Title: Efficacy and Safety of AVE1625 as a Co-treatment With Antipsychotic Therapy in Schizophrenia
Acronym: CONNECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following a pre-specified interim analysis and Data Monitoring Committee recommendation due to insufficient level of efficacy
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6726
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia
Keywords: psychometrics; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — AVE1625

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- AVE1625 dose level 1 (Experimental)
  Interventions: Drug: AVE1625
- AVE1625 dose level 2 (Experimental)
  Interventions: Drug: AVE1625
- AVE1625 dose level 3 (Experimental)
  Interventions: Drug: AVE1625

INTERVENTIONS:
Drug: AVE1625 — oral administration
  Other Names: Drinabant
  Arms: AVE1625 dose level 1; AVE1625 dose level 2; AVE1625 dose level 3
Drug: placebo — oral administration
  Arms: Placebo

SUMMARY:
AVE1625 is a new potent and selective cannabinoid 1 (CB1) antagonist in clinical development for the treatment of cognitive impairment in patients diagnosed with schizophrenia.

The main objective of this study is to evaluate the efficacy on cognitive impairment of 3 doses of AVE1625 using a new cognitive battery called Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) in schizophrenic patients.

The secondary objectives are to measure the efficacy of AVE1625 on functional capacity of the patients using a specific scale called University of California San Diego Performance-based Skills Assessment 2 (UPSA2) and to assess the safety of the compound.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with diagnosis of schizophrenia (diagnosed ≤ 35 years of age).
* Current treatment consisting exclusively of olanzapine, risperidone/paliperidone, quetiapine or aripiprazole monotherapy for at least 2 months.

Exclusion Criteria:

* Inpatient hospitalization within past 3 months.
* Residence at the current address < 3 months due to any instability in the disease.
* Presence of depressive symptoms.
* Past history of clinically significant violent behavior.
* Substance dependence or abuse.
* Pregnant or breast-feeding women or women not protected by effective contraceptive method of birth control.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 873 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the MATRICS Cognitive Battery composite standardized score | at week 24

SECONDARY OUTCOMES:
Change from baseline in the UPSA2 total score | at week 24
Additional scales used for schizophrenia | at week 24
Safety: physical examination, vital signs, ECGs, laboratory parameters, adverse events | study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada

REFERENCES:
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500